CLINICAL TRIAL: NCT02307123
Title: One-year Outcome After Prehospital Intubation
Status: Completed | Type: Observational
Sponsor: Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Toni Pakkanen, MD, MD, Tampere University Hospital
Other Study IDs: 9N088
Record Dates: First submitted 2014-11-30; First posted 2014-12-04 (Estimated); Results first posted 2016-12-22 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2015-12

CONDITIONS: One-year Outcome After Prehospital Intubation
Keywords: Prehospital emergency care (MeSH); Emergency medical services (MeSH); Helicopter emergency medical service, Critical care (MeSH); Airway management (MeSH); Endotracheal intubation (MeSH); Patient outcome
MeSH Terms: interventions — Intubation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HEMS treated patients: Patients whose airways were secured by the HEMS physician.
  Interventions: Procedure: Intubation

INTERVENTIONS:
Procedure: Intubation — HEMS physician prehospital intubation

SUMMARY:
The primary aim of this study was to describe the long-term outcome of critically ill or severely injured patients not in cardiac arrest treated by an EMS physician.

DETAILED DESCRIPTION:
The aim of helicopter emergency medical services (HEMS) is to supplement ground EMS units in the care of prehospital patients. The need for advanced airway management in critical out-of-hospital patients can be considered as one indicator of the severity of the patient's condition.

A recent European initiative suggested advanced airway management to be included in the top five research priorities for physician-provided prehospital care.To our knowledge, no previous studies describe the long-term outcome of critical prehospital patients treated by an EMS physician.

The primary aim of this study was to describe the long-term outcome of critically ill or severely injured patients not in cardiac arrest treated by an EMS physician. Our secondary aims were to determine the indications and causes for EMS physician performed prehospital endotracheal intubation.

ELIGIBILITY:
Inclusion Criteria:

* All non-cardiac arrest patients.

Exclusion Criteria:

* Patients with a known need for personal assistance in activities of daily life prior to the incident leading to prehospital intubation (outcome evaluation).
* Patients intubated by EMS before HEMS arrival.
* Death on scene or during transportation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All non-cardiac arrest patients, whose airway was secured by the HEMS physician.
Sampling Method: Probability Sample
Enrollment: 483 (Actual)
Dates: Start 2013-01; Primary Completion 2014-01 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arvi Yli-Hankala, professor, Study Director — Tampere University Hospital; Toni VS Pakkanen, MD, Principal Investigator — Tampere University Hospital; Ilkka Virkkunen, MD, PhD, Study Chair — Tampere University Hospital; Tom Silfvast, MD, PhD, Study Chair — Helsinki University Central Hospital; Tarja Randell, MD, PhD, Study Chair — Helsinki University Central Hospital

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HEMS Treated Patients
Started | 483
Completed | 483
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | HEMS Treated Patients
Number analyzed (Participants) | 483
Age, Continuous [Median (Full Range); unit: years] | 47.8 [0 to 91]
Gender [Count of Participants; unit: Participants]
  Female | 164
  Male | 319

OUTCOME MEASURES:

1. Primary Outcome: Mortality
Time Frame: 1 year
Measure: Number; unit: percentage of one year mortality
Arm/Group | HEMS Treated Patients
Number analyzed (Participants) | 483
percentage of one year mortality | 35

2. Secondary Outcome: Glasgow Outcome Score (GOS)
Description: GOS 1 = Death GOS 2 = Poor neurological outcome GOS 3 = Good neurological outcome Modified from the original 5 - step classification.
Time Frame: 1 year
Measure: Number; unit: percentage of good neurological outcome
Arm/Group | HEMS Treated Patients
Number analyzed (Participants) | 483
percentage of good neurological outcome | 55

ADVERSE EVENTS:
Arm/Group | HEMS Treated Patients
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No